CLINICAL TRIAL: NCT03004950
Title: Biomarker Effectiveness Analysis in Contrast Nephropathy
Brief Title: Biomarker Effectiveness Analysis in Contrast Nephropathy (BEACON)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Raghavan Murugan, M.D., University of Pittsburgh
Other Study IDs: PRO16090669; R01DK106256-01A1 (NIH)
Record Dates: First submitted 2016-12-23; First posted 2016-12-29 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Acute Renal Failure; Kidney Diseases; Chronic Kidney Disease; Coronary (Artery); Disease
MeSH Terms: conditions — Acute Kidney Injury; Kidney Diseases; Renal Insufficiency, Chronic; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is an observational non-interventional study which will examine a) the accuracy of biomarkers in predicting renal and cardiovascular outcomes after contrast-induced acute kidney injury.

This study will obtain de-identified human plasma & urine samples and corresponding de-identified research study data on subjects who are enrolled into the Prevention of Serious Adverse Events Following Angiography (PRESERVE) study and Biomarker Collection and Analysis in the PRESERVE Trial (VA CSP #578). Biomarker analyses will be performed on the de-identified samples and merged with de-identified research study data.

DETAILED DESCRIPTION:
Contrast-induced acute kidney injury (CIAKI) is a serious complication occurring in patients with chronic kidney disease undergoing angiography and is associated with adverse renal and cardiovascular outcomes. The investigators will address two key questions that remain in high-risk patients undergoing angiography. First, early detection of CIAKI after contrast exposure is problematic because rise in serum creatinine or decline in urine output occur over several days and many cases are under-diagnosed. Second, early risk stratification for long-term adverse events is also problematic because existing risk prediction models only have a modest predictive value. Availability of a biomarker that detects subclinical CIAKI before creatinine and also aids in risk stratification will change primary and secondary prevention strategies. The FDA has recently approved two novel, highly sensitive, urinary cell cycle arrest biomarkers for early detection of AKI. The investigators have shown that these biomarkers: tissue inhibitor of metalloproteinase (TIMP)-2 and insulin growth factor binding protein (IGFBP)7, detect AKI before serum creatinine in critically ill patients and are associated with long-term adverse outcomes. Whether these markers can be used to predict renal and cardiovascular outcomes in patients undergoing angiography is yet unknown. The investigators have been recently funded by the Department of Veterans Affairs to conduct a multicenter, randomized, clinical trial in 7,680 high-risk patients undergoing angiography to compare the effectiveness of intravenous sodium bicarbonate with isotonic sodium chloride, and oral N- acetylcysteine with placebo, for the prevention of serious adverse outcomes associated with CIAKI. The NIDDK has funded an associated biorepository to examine known and yet-to-be identified biomarkers for CIAKI. The investigators propose to leverage these resources to conduct an ancillary observational study entitled Biomarker Effectiveness Analysis in Contrast Nephropathy (BEACON). Using urine and plasma samples obtained before and at four hours after angiography in 1,100 subjects, the investigators will address two specific aims. Aim 1 will examine the accuracy of urinary TIMP-2, IGFBP7, and select other plasma biomarkers in predicting the composite renal outcome of death, dialysis dependence, or persistent renal injury at day 90 after contrast exposure (Aim 1a); biomarker reclassification of risk for adverse renal outcomes and develop a risk score (Aim 1b); and predicting the progression of chronic kidney disease (Aim 1c). Aim 2 will examine the accuracy of urinary TIMP-2 and IGFBP7 in predicting the composite outcome of hospitalization with acute coronary syndrome; heart failure; cerebrovascular accident; or all-cause mortality within 90 days (Aim 2a); and biomarker reclassification of risk for cardiovascular events (Aim 2b). The proposed work will advance NIDDK's mission of early detection, risk-stratification, and prognostication of CIAKI. It will provide new scientific knowledge on using biomarkers to monitor patients undergoing angiography and will have a high impact on clinical practice, physicians, and policy makers.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective or urgent coronary or non-coronary angiography with iodinated contrast media in which it is anticipated that there will be an interval of ≥3 hours between the identification of the indication for angiography and the time of the planned procedure
* Pre-angiography eGFR <60 ml/min/1.73 m2 with diabetes mellitus or pre-angiography eGFR <45 ml/min/1.73 m2 with or without diabetes mellitus
* Ability to provide informed consent

Exclusion Criteria:

* Currently receiving hemodialysis, peritoneal dialysis, continuous renal replacement therapy, or slow low efficiency dialysis
* Stage 5 chronic kidney disease (eGFR <15 mL/min/1.73 m2)
* Unstable baseline serum creatinine (if known) at the time of angiography defined by a change in serum creatinine of ≥25% over the 3 days prior to angiography
* Decompensated heart failure requiring any of the following therapies at the time of angiography
* Emergent angiography procedures defined as an anticipated duration of <3 hours between the identification of the indication for angiography and the time of the planned procedure. We are excluding these patients due to the limited time to collect necessary research data and to ensure that research procedures do not interfere with clinical care
* Receipt of intravascular iodinated contrast within the 7 days preceding angiography
* Receipt of oral or IV NAC within the 48 hours preceding angiography
* Known allergy to NAC
* Known allergy to iodinated contrast media
* Age <18 years
* Pregnancy
* Prisoner
* Ongoing participation in a concurrent interventional study
* Eligible patients who indicate at the time of recruitment an unwillingness to comply with the 96-hour and 90-day outcome assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1,100 men and women enrolled into the PRESERVE trial (NCT01467466)
Sampling Method: Non-Probability Sample
Enrollment: 922 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Predicting the composite renal outcome of death, dialysis dependence, or persistent renal injury, biomarker reclassification of risk for adverse renal outcomes and develop a risk score, and predicting the progression of chronic kidney disease | Day 90 after contrast exposure

SECONDARY OUTCOMES:
urinary biomarkers in predicting the composite outcome of hospitalization with acute coronary syndrome; heart failure; cerebrovascular accident; or all-cause mortality within 90 days, | Within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Raghavan Murugan, MD, MS, FRCP, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murugan R, Boudreaux-Kelly MY, Kellum JA, Palevsky PM, Weisbord S. Contrast-associated acute kidney injury and cardiovascular events: a secondary analysis of the PRESERVE cohort. Clin Kidney J. 2023 Sep 1;16(12):2626-2638. doi: 10.1093/ckj/sfad214. eCollection 2023 Dec. PMID 38046040
- [Result] Murugan R, Boudreaux-Kelly MY, Kellum JA, Palevsky PM, Weisbord S; Biomarker Effectiveness Analysis in Contrast Nephropathy (BEACON) Study Investigators. Kidney Cell Cycle Arrest and Cardiac Biomarkers and Acute Kidney Injury Following Angiography: The Prevention of Serious Adverse Events Following Angiography (PRESERVE) Study. Kidney Med. 2022 Dec 21;5(3):100592. doi: 10.1016/j.xkme.2022.100592. eCollection 2023 Mar. PMID 36874509